CLINICAL TRIAL: NCT06330896
Title: Disease Characteristics and Treatment Response in Plasma Cell Disorders Patients Based on Genetic Abnormalities From Fluorescence In Situ Hybridization and Next Generation Sequencing
Acronym: genetics MM
Status: Not yet recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Chutima Kunacheewa, lecturer, Siriraj Hospital
Other Study IDs: 346/2566(IRB3)
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Plasma Cell Disorder
Keywords: Plasma Cell Disorder; genetic abnormalities; Fluorescence In Situ Hybridization; FISH; Next Generation Sequencing; NGS
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to study the genetic landscape in patients with Plasma Cell Disorders including MGUS, SMM, MM, and amyloidosis in Thailand. The main questions it aims to answer are:

* genetic landscape in patients with Plasma Cell Disorders including MGUS, SMM, MM, and amyloidosis in Thailand who were performed FISH and/or NGS testing
* genetic correlation and genetic dependency between FISH and NGS, stratified by high- and standard-risk groups based on FISH testing in Thai MM patients.
* disease characteristics and response rates in MM patients with cytogenetic abnormalities detected by FISH and/or genetic mutations detected by NGS.
* correlation between cytogenetic abnormalities identified by FISH and genetic mutations detected by NGS with progression-free survival in MM patients.

The FISH and/or NGS testing results, disease characteristics, treatment, and treatment outcomes of patients with plasma cell disorders who underwent FISH and/or NGS testing before IRB approval will be collected through retrospective chart review. Subsequently, data will be gathered prospectively. Participants will provide approximately 12 mL of bone marrow fluid for FISH and NGS testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Plasma Cell Disorders including MGUS, SMM, MM, and amyloidosis
* Aged 18 years and older
* Performed FISH and/or NGS testing
* Has treatment follow up at least one year

Exclusion Criteria:

* Patients with missing crucial data that renders them unanalyzable
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Plasma Cell Disorders including MGUS, SMM, MM, and amyloidosis who were performed FISH and/or NGS testing
Sampling Method: Probability Sample
Enrollment: 498 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
genetic landscape of PCD | 18 months in 498 patients
  number and percentage of genetic landscape of FISH and NGS in patients with Plasma Cell Disorders

SECONDARY OUTCOMES:
genetic correlation | 18 months in MM patients
  genetic landscape correlation between FISH and NGS in MM patients
genetic landscape of relapse MM patients | 18 months in MM patients
  number of genetic landscape in relapse MM patients
overall survival | 18 months
  time of survival in MM patients
progression free survival | 18 months
  time of disease progression in MM patients
factor of genetic landscape differentiation | 18 months in MM patients
  number of MM patients who have the different factors such as gender, age, and comorbidities.
gender | 18 months in 498 patients
  number and percentage of male and female
age | 18 months in 498 patients
  age in years

IPD SHARING:
Plan to Share IPD: Undecided
Need a consensus from colleagues